CLINICAL TRIAL: NCT07195851
Title: Dermatological Safety and Skin Compatibility Evaluation of Test Product Following Cosmetics Europe: Product Test Guidelines for Assessment of Human Skin Compatibility (Colipa Standard, 1997)
Brief Title: Dermatological Safety and Skin Compatibility Evaluation of Test Products
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: OneSto Labs Private Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB250039-OL
Record Dates: First submitted 2025-09-16; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Each participant will receive test products patches on the forearm, including the test product(s), a negative control (0.9% Saline), and a positive control (1% sodium lauryl sulfate).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm includes 4 test products along with positive and negative control (Experimental): Below interventions along with 1% SLS (Positive control) and 0.9% Normal saline (Negative Control) will be applied in subject's forearm
  1. Bare Anatomy Expert Advanced Hair Growth Serum
  2. Bare Anatomy Expert Ultra-Smoothing Shampoo
  3. Bare Anatomy Expert Ultra-Smoothing Hair Serum
  4. Bare Anatomy Expert Ultra-Smoothing Hair Mask
  Interventions: Other: 1.Bare Anatomy Expert Advanced Hair Growth Serum 2.Bare Anatomy Expert Ultra-Smoothing Shampoo 3.Bare Anatomy Expert Ultra-Smoothing Hair Serum 4.Bare Anatomy Expert Ultra-Smoothing Hair Mask

INTERVENTIONS:
Other: 1.Bare Anatomy Expert Advanced Hair Growth Serum 2.Bare Anatomy Expert Ultra-Smoothing Shampoo 3.Bare Anatomy Expert Ultra-Smoothing Hair Serum 4.Bare Anatomy Expert Ultra-Smoothing Hair Mask — Dose: 0.1 ml of sample solution Route of administration: Topical Mode of usage: Products will be evaluated through the complete occlusion for 48 hours.

SUMMARY:
Dermatological Safety and Skin Compatibility Evaluation of Test Product following Cosmetics Europe: Product Test Guidelines for Assessment of Human Skin Compatibility (Colipa Standard, 1997)

DETAILED DESCRIPTION:
This is single-centre, evaluator blinded study in healthy human subjects. single 48-hour application of sponsors provided test product along with positive and negative control will be kept in contact with the skin for at least 48hours (± 2hours).safety will be assessed through the study by monitoring of adverse event. A sufficient number 26 subject will be enrolled to get 24 to complete the study. There are total four visits in this study. Visit 01 (Day01):Screening, Enrolment and Patch Application, Visit 02 (Day 03):Patch Removal & 30 ± 5 min irritation scoring upon patch removal. Visit 03 (Day 04): 24 (± 2 hour)irritation scoring (Day 04)Visit 05:

At 48±2 hours Irritation Scoring

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years (both inclusive) at the time of consent.
2. Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
3. Subject with normal Fitzpatrick skin type III to VI (Human skin colour determination scale).
4. Females of childbearing potential must have a self-reported negative pregnancy test.
5. Subject who do not have any previous history of adverse skin conditions and are not under any medication likely to interfere with the results.
6. Subject is in good general health as determined by the Investigator on the basis of medical history.
7. Subjects is willing to maintain the test patches in designated positions for 24 Hours.
8. Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
9. Subject must be able to understand and provide written informed consent to participate in the study.
10. Subject is willing to refrain from vigorous physical exercise during the study period and follow all the instruction given.
11. For Sensitive Specific Skin Study Only:

    * Subject scoring greater than 30 for Section 2 - Sensitive v/s Resistant skin in modified Dr Baumann's skin type questionnaire.
    * Subject with sensitive skin as confirmed by Lactic Acid stinging test.

Exclusion Criteria:

1. Subject having skin irritation, blemishes, excessive hair, moles, pigmentation, pimples, marks (e.g. tattoos (within the previous 3 months), scars, sunburn), open wounds, cuts, abrasions, irritation symptoms or any dermatological condition on the test site(s) i.e. back that can interfere with the reading.
2. Medication which may affect skin response and/or past medical history.
3. Subject having history of diabetes
4. Subject have history of mastectomy for cancer involving removal of lymph nodes within the past year, or treatment of any type of cancer within the last 6 months.
5. Subject suffering from any active clinically significant skin diseases which may contraindicate.
6. Subject having history of any skin diseases including eczema, atopic dermatitis or active cancer.
7. Participation in any patch test for irritation or sensitization within the last four weeks.
8. Subject having history of asthma or COPD (Chronic obstructive pulmonary disease).
9. Use of any:

   i. Prescribed or over-the-counter (OTC) anti-inflammatory drug within five (5) days prior to application. ii. Antihistamine medication or immunosuppressive drugs within seven (7) days prior to first patch application. iii. Systemic or topical corticosteroids at patch site within four (4) weeks of test product application (steroidal nose drops and/or eye drops are permitted)
10. Topical drugs used at application site.
11. Subject with Self-reported Immunological disorders such as HIV positive, AIDS and/or systemic lupus erythematous.
12. Individual who has a medical condition or is taking or has taken a medication which, in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk.
13. Subject with known allergy or sensitization to medical adhesives, bandages.
14. Participation in other patch study simultaneously.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the dermatological safety of the test products assessed by 48-hour patch test under complete occlusion condition. | 30 ± 5 minutes post patch removal (Day 03), 24 ± 2 hours post patch removal (Day 04), and 48 ± 2 hours post patch removal (Day 05).
  Dermatological reactions will be evaluated using the 48-hour patch test method under complete occlusion. Assessments will be performed to detect any skin irritation, erythema, or other local reactions at the application site.

SECONDARY OUTCOMES:
Skin Safety Evaluation by assessing Change in Transepidermal Water Loss (TEWL) at the Application Site | at baseline, 30 mins and 24 hours post patch removal
  Transepidermal Water Loss (TEWL) at the site of product application will be measured using the TEWAMeter TM Hex to assess the impact of the investigational product on skin barrier function

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan Patel, Principal Investigator — NovoBliss Research Private Limited

IPD SHARING:
Plan to Share IPD: No